CLINICAL TRIAL: NCT00585741
Title: Pilot Study of 18F-FLT Pet Imaging in Cancer Patients
Brief Title: Pilot Study of 18F-FLT PET
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-2006-0280
Record Dates: First submitted 2007-12-21; First posted 2008-01-03 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: CNS Brain Metastasis; Head and Neck Cancer; Lung Cancer; Prostate Cancer; Esophageal Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Esophageal Neoplasms | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 2. Head and neck (Experimental): Imaging with 18F-FLT PET
  Interventions: Procedure: Imaging with 18F-FLT PET
- 3. Lung (Experimental): Imaging with 18F-FLT PET
  Interventions: Procedure: Imaging with 18F-FLT PET
- 4. prostate (Experimental): Imaging with 18F-FLT PET
  Interventions: Procedure: Imaging with 18F-FLT PET
- 5. esophagus (Experimental): Imaging with 18F-FLT PET
  Interventions: Procedure: Imaging with 18F-FLT PET
- 1.CNS (Experimental): Imaging with 18F-FLT PET
  Interventions: Procedure: Imaging with 18F-FLT PET

INTERVENTIONS:
Procedure: Imaging with 18F-FLT PET — Imaging with 18F-FLT PET
  Arms: 1.CNS
Procedure: Imaging with 18F-FLT PET — Imaging with 18F-FLT PET
  Arms: 2. Head and neck
Procedure: Imaging with 18F-FLT PET — Imaging with 18F-FLT PET
  Arms: 3. Lung
Procedure: Imaging with 18F-FLT PET — Imaging with 18F-FLT PET
  Arms: 4. prostate
Procedure: Imaging with 18F-FLT PET — Imaging with 18F-FLT PET
  Arms: 5. esophagus

SUMMARY:
Fractionated radiotherapy induces an observable change in the proliferative activity as assessed by pre-treatment and early-treatment 18F-FLT PET imaging. This study is designed to investigate 18F-FLT as a PET imaging agent for predicting treatment effectiveness in several tumors and will serve as a pilot study to a planned PO1 submission

ELIGIBILITY:
Inclusion Criteria:

* Able to tolerate a PET/CT scan
* Age of 18 or older
* signed informed consent
* being considered for radiotherapy for treatment of CNS mets, Head and neck cancer, lung cancer, prostate cancer or esophageal cancer

Exclusion Criteria:

* Prior XRT to site being studied
* severe claustrophobia or inability to tolerate PET/CT
* unable to provide written consent
* pregnant or breastfeeding women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To test whether the cellular response to fractionated radiotherapy leads to observable global change in the uptake of 18F-FLT as assessed by PET imaging | end of study

SECONDARY OUTCOMES:
To assess the technical and logistic feasibility of 18F-FLT scans in a population of cancer patients | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jeraj, Ph.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and clinis, Madison, Wisconsin, United States